CLINICAL TRIAL: NCT04199130
Title: Effectiveness of Combined Attention and Metacognitive-strategy Training Approaches to Cognitive Impairment in Moderate-to-severe TBI
Brief Title: Cognitive Rehabilitation and Brain Activity of Attention-Control Impairment in TBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed with the IRB due to slow enrollment during COVID. Will be modifying the study with a new submission.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201902218
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Described in study description
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Experimental): This arm will receive BrainHQ for the first four weeks of the study, and Goal Management Training for the second four weeks.
  Interventions: Behavioral: BrainHQ; Behavioral: Goal Management Training
- Intervention Group 2 (Experimental): This arm will receive Goal Management Training for the first four weeks of the study, and BrainHQ for the second four weeks.
  Interventions: Behavioral: BrainHQ; Behavioral: Goal Management Training
- Treatment-as-usual (No Intervention)

INTERVENTIONS:
Behavioral: BrainHQ — BrainHQ is a web-based "brain-training" program. The investigators will assign participants to attention specific modules that they will complete at home with the goal of "restoring" attentional functions lost through injury via repetitive tasks of graded difficulty.
  Arms: Intervention Group 1; Intervention Group 2
Behavioral: Goal Management Training — This is a manualized, interactive, metacognitive-strategy training designed to promote a mindful approach to complex real-life tasks and reduce lapses in attention via implementation of "compensatory" mechanisms for monitoring tasks.
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
The purpose of this research study is to develop a method to improve thinking difficulties in individuals who have experienced a traumatic brain injury and report experiencing difficulties in attention and concentration. This study aims to understand how cognitive rehabilitation of attention difficulties affects brain activity.

DETAILED DESCRIPTION:
This study will compare the effectiveness of two different types of cognitive rehabilitation in moderate-to-severe (m/s) traumatic brain injury (TBI) survivors. More specifically comparisons will be made between Direct Attention Training administered via BrainHQ, and Metacognitive Strategy Training in the form of the evidence-based Goal Management Training (GMT) protocol.

These interventions will be compared to the standard of care, to each other, and their combined effectiveness will be assessed. Groups will consist of randomized individuals with moderate-to-severe TBIs who experience attention deficits. Each treatment will be administered for 4 weeks and two intervention groups will be used to counterbalance treatment order. Group 1 will receive BrainHQ first followed by GMT, while Group 2 will receive GMT first followed by BrainHQ. In addition a third group will serve as a treatment-as-usual control group.

Primary outcomes include measures of self-care, ability, adjustment and participation. Secondary outcomes include measures of cognition and brain function. And lastly, tertiary outcomes include measures of emotional and psychosocial functioning. These outcomes will be measures at baseline, following completion of the first 4 week treatment in both groups (Group 1 = BrainHQ while Group 2 = GMT), and following completion of the second 4 week treatment in both groups (Group 1 = GMT while Group 2 = BrainHQ).

ELIGIBILITY:
Inclusion Criteria:

* Self-report of attention problems, confirmed with psychometric testing
* Ruff 2 & 7 selective attention task score ≤ 1.5 standard deviations from demographically-matched norms
* Able to participate in study at 12-60 months post-injury without contraindications
* Willingness to be randomized and to participate in treatment procedures
* Capacity to visit the laboratory for repeated treatment sessions and testing
* Access to internet-enabled home computer
* English as native language
* Adequate reading comprehension to allow completion of questionnaires
* Reliable digit span (RDS) score > 7

Exclusion Criteria:

* Pre-existing neurological disorder associated with cerebral dysfunction (e.g., stroke, history of epilepsy or chronic seizure disorder)
* Current alcohol or drug use
* Pre-existing severe psychiatric disorder (e.g., schizophrenia) detected by Mental Screening form, 3rd edition (MHS-III) or history of psychiatric diagnosis sufficiently severe to have resulted in inpatient hospitalization
* Current suicidal/homicidal ideation or intent
* Reported involvement in current litigation
* Reported history of pre-injury learning disability
* Not competent to provide written informed consent (i.e., not able to demonstrate understanding or expectations of study and potential risks of participation)
* Does not fully understand the nature of the study and requirements of participation
* Does not understand task instructions
* Validity testing (score ≤ 7) on the RDS 22 test of suboptimal/non-credible performance taken from the forward and backward digit span subtests of the WAIS-IV

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Measurement of change in self-care | Measured at Baseline, Post treatment 1 (4 weeks post-baseline), Post treatment 2 (8 weeks post baseline)
  These will be measured via the Timed Instrumental Activities of Daily Living assessment. Participants will be timed performing common functional tasks and longer completion times indicate greater impairment.
Measurement of change in ability, adjustment and participation | Measured at Baseline, Post treatment 1 (4 weeks post-baseline), Post treatment 2 (8 weeks post baseline)
  A composite self-report questionnaire known as the Mayo-Portland Adaptability Inventory will be used to measure functioning across these domains. This measures uses a scale from 0 to 4. The higher the score the more severe the impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Public Health and Health Professions, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No